CLINICAL TRIAL: NCT06311188
Title: Exploring PTSD Symptoms, Barriers and Facilitators to Mindfulness-based Stress Reduction for Justice-Involved Black/African American Female Adolescents and Parents/Caregivers
Brief Title: Exploring PTSD Symptoms, Barriers and Facilitators to Mindfulness
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Camille Renee' Quinn, Associate Professor of Social Work, School of Social Work, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00240243; 1R21MD016940-01A1 (NIH)
Record Dates: First submitted 2024-02-22; First posted 2024-03-15 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Stress; Trauma; PTSD; HPA
Keywords: Nonrandomized trial; Black girls; Legal system involvement; Cortisol Biomarker
MeSH Terms: conditions — Wounds and Injuries; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Single arm trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ITR Healing Intervention (Experimental): This is a single arm nonrandomized test of the culturally adapted ITR healing intervention.
  Interventions: Behavioral: ITR Healing intervention

INTERVENTIONS:
Behavioral: ITR Healing intervention — This is a nonrandomized test of the culturally adapted ITR healing intervention that is based on the ITR framework. The ITR Healing intervention comprises six 60-minute sessions based on Intersectionality theoretical framework, Healing Centered Engagement (HCE) activities that were integrated into the intervention, as well as participant's feedback about the intervention. Also, the participants' behavioral experiences per the Theoretical Domains Framework targets was used to adapt the intervention activities. HCE focuses on building a holistic approach and empathy for each session, i.e., using music, dance/movement, meditation, breathing and journaling.

SUMMARY:
The purpose of this study is to investigate justice-involved Black/African American female adolescents' (JI BAFAs; N=35) self-reported outcomes: stress, posttraumatic stress disorder (PTSD), recidivism, etc., as well as their parents/caregivers' (P/Cs; N=35) stress and pre- and post- intervention results along with their views of an adapted intervention.

DETAILED DESCRIPTION:
This study was conceptualized via an initial partnership with the Principal Investigator (PI), the City of Columbus Commission on Black Girls (Commission or COBG) and the Franklin County Juvenile Court. The investigators will also conduct individual semi-structured interviews with providers (N=20) to assess their views of the adapted intervention, as well as who they think will be best to deliver the intervention, and in which settings/locations. Further, the investigators will create three advisory boards: Community Advisory Board, Scientific Advisory Board, and a Youth Advisory Board to assist the research team with recruitment, study design and implementation, intervention development, and to ensure the rigor and translational aspects of the research study. The investigators will use all the identified themes from the JI BAFA, P/C, and provider interviews to adapt and test a healing centered stress reduction intervention for Phase II of the study. The investigators will recruit JI BAFA-P/C dyads for Phase II of the study and Phase I participants will be invited to participate.

The objectives of this research study are to:

1. Assess JI BAFAs' PTSD, as well as their and their P/Cs' stress.
2. Culturally adapt a healing centered stress reduction intervention based on the responses from ten JI BAFA-P/C dyads, including ten Black girls ages 14-18 who are involved with the Franklin County Juvenile Court and ten of their parents/caregivers based on their feedback to identify specific gaps in service provision and utilization of services, i.e. barriers to treatment, as well as describe the proposed intervention and elicit their feedback about its utility and implementation. Intervention development and adaptation will also be based on the feedback from 20 providers, and recommendations from select advisory board members.
3. Test the culturally adapted intervention and assess the participants' experiences via member checking, a method used to ensure the accuracy of what they told us in the interviews at the end of the interview.
4. Identify specific gaps in service provision and utilization of services.
5. Provide recommendations to study participants and Franklin County Juvenile Court to inform practice protocols, and a future randomized control trial to test this culturally adapted intervention with a larger sample of participants.

ELIGIBILITY:
Inclusion Criteria:

* Black girls aged 14-18
* Black girls with a misdemeanor and/or felony charge in their lifetime
* Positive PTSD screen (PC-PTSD score of 2 or more; if more than one JI BAFA are from the same family, the investigators will recruit the girl with the highest PTSD score)
* Black girls report juvenile justice involvement within 12 months prior
* Black girls live with a P/C (mothers, fathers, and other caregivers/legal guardians) who will also participate in the study
* Parents/Caregivers nominated by the girls to participate in the study who are between the ages of 18 and 90 years of age
* Legal/ social services providers / educators who work with the population.

Exclusion Criteria:

* Prisoners per the IRB definition
* Black girls who are younger than 14 and older than 18
* Severe cognitive delay so the youth cannot complete the assessment instruments, as measured using the Montreal Cognitive Assessment (MoCA)
* Active psychosis requiring a greater level of care [Structured Clinical Interview for DSM Disorders (SCID)]. Screening for the study will take place prior to consent/assent of the study participants
* Parents/Caregivers who are not nominated by the girls to participate in the study who are not between the ages of 18 and 90 years of age
* Legal/ social services providers / educators who have been working with the population for less than three years.

Ages: 14 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self representation and self disclosure of their gender.
Enrollment: 90 (Estimated)
Dates: Start 2026-01-08 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
PTSD Screen | 24 months
  PTSD psychiatric disorder that may occur in people who have experienced or witnessed a traumatic event such as a natural disaster, a serious accident, a terrorist act, war/combat, or rape or who have been threatened with death, sexual violence or serious injury. PTSD Will be measured by the Primary Care PTSD Screen, which all participants will complete. . The authors suggest that in most circumstances the results of the PC-PTSD should
  Those screening positive should then be assessed with a structured interview for PTSD. The screen does not include a list of potentially traumatic events.
PTSD Checklist | 24 months
  PTSD Checklist from DSM-5 (PCL-5), which all participants will complete. A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items.

SECONDARY OUTCOMES:
Stress Psychosocial | 24 months
  Perceived Stress Scale Questionnaire-short, 10 items. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Stress Physiological | 24 months
  Hair assessment and provide 1-3 cm of hair will be assessed via enzyme-linked immunosorbent assay at the Ford Stress Science Lab for mean cortisol. Hair will be cut from the posterior vertex of the scalp. Ideally participants will have 3 cm of hair for assay but if they have 1 cm will be included to avoid selection bias; hair length can be included as a covariate in analysis if needed. Participants will be screened on hair care practices (chemical use, shampoo frequency), medications (steroids, estrogen/progesterone) to assess the effect on cortisol. The hair cortisol captures cumulative exposure to cortisol over time as each 1 cm of hair growth approximates 1 month of mean cortisol output.
Parent/Caregiver-Child Relationship | 24 months
  All participants will complete a 4-item Parent/Caregiver-Child Relationship Scale to assess the quality of their relationships. These items will be reverse scored so that a lower score indicates less of a relationship and a higher score indicates more of a relationship.
Five Facet Mindfulness Questionnaire (FFMQ) | 24 months
  FFMQ assesses actions, non-judgmental inner experience, and non-reactivity. Direct Scoring with Likert values and higher scores are indicative of someone who is more mindful in their everyday life.
Recidivism | 24 months
  Delinquency Scale 2 questions with 16 items. If none are selected, the minimum is 0 and the maximum selected is 16.
Personal Agency | 24 months
  Only adolescent girls will complete 6-item Personal Efficacy Scale that measures the youth's perception of their ability to solve problems and perform jobs well. Maximum score is 6 and the minimum score is 1, with higher scores considered more and lower scores considered less.
Racial Identity | 24 months
  Only adolescent girls will complete the centrality subscale of the Multidimensional Inventory of Black Identity (MIBI) to measure racial identity. The minimum score would be 8 and maximum score would be 24 with the higher score noting more and the lower score noting less racial centrality.
Parenting Stress | 24 months
  Parenting Stress Questionnaire-short. Only parents/caregivers will complete the 18-item. A low score signifies a low level of stress, and a high score to signifies a high level of stress.

OTHER OUTCOMES:
MoCA screen | 20 months
  Everyone interested in participating in the study will complete the Montreal Cognitive Assessment - one of three screeners for study eligibility. The maximum score is 30 and the minimum score is 1.
CESD - Depression screen | 20 months
  Everyone interested in participating in the study will complete the Center for Epidemiologic Studies Depression Scale to screen for depression, wth internal consistency = .85-.90.
  MBSR has been effectively modified for depressed individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Power-Carter, PhD, Study Director — Ohio State University

IPD SHARING:
Plan to Share IPD: Yes
Sharing of data generated by this project is an essential part of our proposed activities and will be carried out in several different ways. The investigators wish to make our results available to the community of scientists and the planning and community-based organizations and other organizations serving young Black youth. Conversely, the investigators welcome collaboration with others who could make use of the protocols developed in the project. The investigators will share results from surveys and interview data after de-identification through the Inter- University Consortium for Political and Social Research (ICPSR), an NIH funded data repository, within one year of completion of data collection (see https://www.icpsr.umich.edu/icpsrweb/). Submitted data will conform with relevant data and terminology standards.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The investigators agree to deposit data into ICPSR repository as soon as possible but no later than within one year of the completion of the funded project period for the parent award or upon acceptance of the data for publication, or public disclosure of a submitted patent application, whichever is earlier.
Access Criteria: Members of ICPSR will be able to access our deidentified data per their eligibility requirements.
URL: https://www.icpsr.umich.edu/icpsrweb/